CLINICAL TRIAL: NCT01326832
Title: Prospective Study for Evaluation of Proximally Anchored (Metaphysis) Cementless Femoral Component for Total Hip Arthroplasty. 10 Year Clinical Evaluation,DXA and RSA Follow-up of Primoris® Femoral Component.
Brief Title: 10 Year Clinical Evaluation of Primoris Hip Component
Acronym: Primoris
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet Denmark A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BMETEU.CR.UK4A
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Coxarthrosis
Keywords: THA
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primoris: 50 patients included in RSA cohort of total of 350 anticipated Primoris cases
  Interventions: Device: Primoris

INTERVENTIONS:
Device: Primoris — Total hip arthroplasty with the new Primoris femoral component

SUMMARY:
Using the traditional and hitherto used uncemented hip prostheses achieved good clinical results, but one of the drawbacks is the risk of fracture in the femoral shaft in indbankning of the prosthesis (1-2%). In addition, the bone scan demonstrated that in the years after surgery dropped almost 30% of bone mass in the femoral shaft. This bone loss increases the risk that in the years after surgery, the increased risk of fractures around the prosthesis and in addition to impeding the described bone replacement prosthesis later.

The newly developed prosthesis is anchored in the femoral neck and thus not involve the femoral shaft. This ensures a more physiological or normal weight transfer to the femur bone.

This contributes to bone mass in long large extent preserved in the years after surgery, so you have a better opportunity later to make a new prosthesis surgery with good results. The new prosthesis should be capable of simultaneously reducing the incidence of thigh pain in the first year after surgery.'

DETAILED DESCRIPTION:
By insertion of artificial hip joints in young and middle aged are often used so-called uncemented technique in which the prosthesis is fixed to the bone without the use of bone cement. Anchoring happens when the bone cells grow into the prosthesis porous surface, thereby creating a stable anchorage of the prosthesis, both short and long term.

A hip prosthesis consists of 3 main elements:

1. socket
2. ball
3. femoral component, which hold ball. Femoral component is anchored to the upper end of the femur including the upper 12-15 cm of the marrow cavity.

Achieved good results with this principle. The method involves a risk of fracture at the top end of the femur bone during and after insertion of the prosthesis, but also that there is some bone loss in the year after surgery. Finally there is a 3-10% chance that you get thigh pain due to different elasticity of the femur and the long shank prosthesis.

Based on the foregoing disadvantages of the femoral components, which are commonly used, has for years been experimenting with the introduction of shorter implants, which are either anchored in the femoral neck or femoral neck combined with the very top end of the femur bone (metaphysis). By using such a prosthesis, it is proven to preserve the bone in the upper femur forward and avoids the disadvantage in terms of the above described femoral pain. There is also described problems by using these short prostheses, especially in the form of solution, and pain secondary to anchor bolts in the upper femur forward.

In Orthopaedic Surgery, Region Nordjylland, one has in the period 1999 to 2003 33 such prostheses implanted at clinics in Farsø and Frederikshavn and achieved good results apart from pain similar to the above anchoring screws. At follow-up of these prostheses, using DEXA scans, the investigators have shown that prosthesis, bone-saving, since bone mass at the femoral neck and the very top end of the femur bone is preserved.

From our experience with the aforementioned short prosthesis, the investigators have joined with Biomechanical Institute, Royal National Orthopaedic Hospital, Stanmore, London and firm Biomet developed a modern design of the above. This is a short prosthesis that is anchored in the femoral neck and the upper end of the femur (metaphysis). Prosthesis made of titanium with a porous surface (Bonemaster ®). The prosthesis is anchored during surgery by pressure-fit (press-fit) and in a few weeks the bone grows into the prosthesis.

Prosthesis manufactured in 5 sizes and design of the prosthesis is aligned with a series of CT scans of the femur was carried out at Stanmore in London. Has developed instruments to ensure a uniform instrumentation and minimizing the risk of fractures in connection with the operation. Performed a series of laboratory tests and these tests, the prosthesis was found to be completely stable and even full load stable and the risk of fracture related to prosthesis insertion is minimized.

The current study intends to examine whether that can be achieved equally good clinical results as with the conventional uncemented femoral component and bone mass in the upper end of the femur bone is preserved. Using a specific X-ray analysis (RSA) also assessed the stability between the prosthesis and bone. Both DEXA scan as RSA studies have routine examinations by Orthopaedic Surgery, Region Nordjylland, Klinik Farsø.

The planned surgery 50 young men and women with primary or secondary osteoarthritis of the hip joint. Patients fulfilling the inclusion criteria and not subject to exclusion criteria received oral and written information about the investigation.

Accept the patient to cooperate with the investigation confirmed that the patient's signature approx. 2 weeks after oral and written information is given.

The operation is performed after the usual principles with rear access to the hip joint, removal of rod ends and the insertion of an uncemented socket. After preparing the femoral neck and top of thigh to the insertion of the short femur prosthesis and make selection using tantalumkugler for RSA analysis. When the prosthesis is inserted carried out sample-space theorem and using a 36 mm Co-Cr-ball, which is currently the department's practices. After surgery the patient allowed partial load the first 6 weeks. There is an ongoing clinical and radiographic controls and registration of unforeseen events arising from the use of the product.

If the flow after 2 years are fully comparable clinical outcomes, minimal migration as measured by RSA and final preservation of the bone around the implant, then the use of the implant extends to several clinics at home and abroad, as per the recommendations of the Danish Orthopaedic Association reference program for hip replacement surgery.

When implementing any new implant designs is a lower risk of unforeseen complications in the form of fracture encountered in denture-deployment and subsequent unexpected prosthetic solution. If the burst occurs Intraoperative, you can convert to the deployment of conventional hip prosthesis without involving major risks for the patient. Early prosthetic solution is also possible deployment of conventional complete dentures without result deteriorates. The disadvantages of the possible complications are in the worst case of operation (revision).

In addition, the disadvantages of trial participation increased radiation dose due to 4 additional X-ray checks in the first 2 years after surgery and 4 extra bone scans (DEXA).

The described investigation will clarify whether the theoretical advantages that have hitherto been demonstrated by clinical and biomechanical study (normal weight transfer, bone sparing and bone-keeping in the short and long term), also obtained by applying the newly developed prosthetic component. If so, there will then be able to especially younger patients with osteoarthritis of the hip joints better chance of achieving good clinical outcomes and long-term sustainability by eventual replacement surgery, typically 10-20 years after primary surgery.

Disadvantages of the described study estimated minimal compared to the benefits that a large group of patients could benefit.

The actual cost of conducting the survey shall be borne by the prosthesis manufacturer Biomet UK Ltd.. and Orthopaedic Surgery, North Jutland and the amount transferred to specific research account affiliated research unit of Orthopaedic Surgery, Region Nordjylland and paid through the Budget and Finance, Region House, Region Nordjylland.

ELIGIBILITY:
Inclusion Criteria:

* younger OA patients with good bonestock

Exclusion Criteria:

1. Patients who do not understand the given information to patients
2. Competing disorder requiring treatment with anti-inflammatory drugs (NSAIDs, steroids, cytostatics).
3. Estimated remaining life expectancy < 10 years
4. Rheumatoid arthritis or other arthritis (eg psoriatic arthritis).
5. Previous surgery on relevant hip.
6. Pain Normative and disabling osteoarthritis of the ipsilateral knee.
7. Co-mobiditet (ASA-group 3-5).
8. Neurological disorder which compromises the motor skills and rehabilitation courses.
9. Pregnancy.
10. Osteoarthritis secondary to Calvé-Legg-Perthes' disease and juvenile epifysiolysis coxae.
11. Acetabular dysplasia and secondary subluxation (Crowie grade II to IV).
12. Previously established osteoporosis or osteoporosis detected by current DEXA scan.
13. Ongoing treatment with osteoporosis medications (calcium and vitamin D, bisphosphonates, estrogen receptor modulating agents and parathyroid hormone, etc.).
14. Aseptic caputnekrosis (post-traumatic, idiopathic).
15. Deform the femoral neck (femoral length, measured medially ≤ 15 mm)
16. Varus or valgus deformity in proximal femur inc. femoral (Collum angel < 125 ° or > 145 °.)
17. Retroversion or anteversion femur.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: younger patients with coxarthrosis
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2011-09; Primary Completion 2022-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
RSA | 2 years
  radio stereographic analysis for prosthesis migration

SECONDARY OUTCOMES:
Harris Hip score | 10 years
  Harris Hip score, Harris Hip Score, 0-100 points. The higher the positive difference between baseline and follow up the better the result.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 10 years
  Womac has 3 subscales: Pain score range 0-20, Stiffness score range 0-8, Physical Function score range 0-68. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Poul T NIELSEN, PhD, Principal Investigator — Aalborg University Hospital
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Veijle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Undecided